CLINICAL TRIAL: NCT03782597
Title: Representations and Strategies of Families Faced With Radicalisation Process of Their Young People
Brief Title: Representations and Strategies of Families Faced With Radicalisation Process
Acronym: FamRad
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Institut Mutualiste Montsouris (Other)
Responsible Party: Sponsor
Other Study IDs: PSY-02-2018
Record Dates: First submitted 2018-07-31; First posted 2018-12-20 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Family Members; Adolescent Problem Behavior; Qualitative Research; Young Adult
Keywords: Radicalization

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Semi-structured interviews or focus groups to explore families representations and strategies about their teenagers involved in radicalisation process — A sample of representative French families (parents, siblings, and persons identified as attachment figures) of adolescents or young adults (12-25 years old) involved in the radicalisation process will be asked to participate in semi-structured interviews or focus groups to explore their representations and strategies about radicalisation. It will be supplemented by genogram draw sociodemographic data.

SUMMARY:
Objectives:

This study aims to explore families' representations and strategies about their teenagers or young adults involved in the radicalisation process and use these findings to build specific tools to help professionals provide family support.

DETAILED DESCRIPTION:
Background:

With repeated attacks, literature about radicalization is growing up. But only few have families as concern, whereas during adolescent process, the place of family remains central. Moreover, professionals of health care and social work lack of understanding and specific tools so as to support families.

After the 11th of September, 2001, literature research about terrorism increased by 300%. Many aspects have been investigated. A recent sytematic review studied the early process, pathway and determinant of radicalization and extremism among muslim society. Many themes are described by studies : role of identity, social drivers, individual factors health and personality, precipitating factors, personal experiences, media and government influence, grievances, perpetuating factors, in-group qualities, methods of persuasion. But none of the studies focus on families of radicalized people.

Another recent review explores the radicalization's motivation and links with psychopathology. None study speaks about families; neither to support nor to prevent from radicalisation. In contrast, if families are missing in the study of radicalisation process they appear in "deradicalization process": for self-preservation aim; for grant of pardon and sign of strong attachment; as way to restor self-preoccupation, opposed to radicalization preoccupation. It conclude with importance of social connection to support out of radicalism process in which family and closed community are central and first mentioned.

Besides, family is often at the forefront to realize first breakdowns with currently environment, changes, new friendship and group affiliations. Knowing family sociocultural references of the radicalized people by inside, their views and explanation are very precious; especially when there is subculture or migration history, where parentality, for example isn't thought with the same way according to different origin culture. Moreover in French context, most of the radicalized people are young people: from 15 to 30 years old, with two third between 15 and 21 years old. And during all adolescent process, family role remain central to reach adulthood with inside security enough, supporting autonomisation-separation process.

Among heterogeneity of adolescent and timing process, scientific literature agree that adolescence can happen between 10 and 25 years old. Thus in this period, radicalisation process and recovery can't be understood without view of close entourage (and especially parents or attachment figures).

We found only found a very few studies on families of radicalized people, that don't totally cover the field we will explore, and with no qualitative guidelines criteria reported (COREQ 32).

Methods and Analysis This study aims to explore families' representations and strategies about their teenagers or young adults involved in the radicalisation process and use these findings to build specific tools to help professionals provide family support.

This is a qualitative study supplemented by quantitative data. A sample of representative French families (parents, siblings, and persons identified as attachment figures) of adolescents or young adults (12-25 years old) involved in the radicalisation process will be asked to participate in semi-structured interviews or focus groups to explore their representations and strategies about radicalisation. It will be supplemented by genogram draw and sociodemographic data.

Data will be coded and analysed in accordance with the principles of interpretative phenomenological analysis (IPA), with Nvivo software, and then discussed with the entire research group. At the end, feedback from participants will be sought to ensure the validity of results and obtain their opinion about whether their meanings and perspectives are presented.

The study and the report will follow the COREQ recommendations. After the data are collected and analysed, the tools will be built and tested, before dissemination.

ELIGIBILITY:
Inclusion Criteria:

* Immediate or extended family or "attachment figure" of a person aged 12-25 years who has been convicted of AMP or AT or reported by a family member or professional
* Voluntary consent to participate for adults, and voluntary consent by both minors and their parents or legal guardian.

Exclusion Criteria:

* Immediate or extended family or attachment figure of a young person from 12 to 25 years old,
* reported by a family member or professional (e.g., in health care, social work, teaching, or the court system) for a radicalisation issue to: either the CNAPR or police or a public prosecutor or juvenile court judge, for whom the report did not lead to an inquiry by the DGSI and/or a specific referral (for example, for social work with the PJJ or the Child Welfare department, or for assistance from a healthcare facility, association or a "referent laïcité et citoyenneté"

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A sample of representative French families (parents, siblings, and persons identified as attachment figures) of adolescents or young adults (12-25 years old) involved in the radicalisation process will be asked to participate in semi-structured interviews or focus groups to explore their representations and strategies about radicalisation
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Representations of families | 3 years
  Representations of families face with radicalization process of their adolescent or young people assessed through analysis of face-to-face semi-structured interview with IPA (Interpretative Phenomenological analysis), including descriptive, analytic and synthetic levels of analysis

SECONDARY OUTCOMES:
Strategies of families | 3 years
  Stratégies of families face with radicalization process of their adolescent or young people assessed through analysis of face-to-face semi-structured interview with IPA (Interpretative Phenomenological analysis), including descriptive, analytic and synthetic levels of analysis

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Aude PIOT, MD, PhD, Principal Investigator — Institut Mutualiste Montsouris
Locations (1):
- Adolescents House, Universitary Hospital Cochin, Paris, Île-de-France Region, France